CLINICAL TRIAL: NCT01544712
Title: Treatment of Stage 3 Osteonecrosis of the Femoral Head by Autologous Transplantation of Bone Marrow Cells: a Randomized, Controlled Double Blind Study
Brief Title: Controlled Study of Stage 3 Osteonecrosis Treatment by Bone Marrow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean-Philippe Hauzeur, Principal investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ref 2004/08 st 3
Record Dates: First submitted 2012-02-22; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-02

CONDITIONS: Non Traumatic Osteonecrosis of the Femoral Head (Hip)
Keywords: osteonecrosis; cell-based therapy; bone marrow; mesenchymal stem cell; hip; core decompression
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Core decompression
  Interventions: Procedure: core decompression of the femoral head
- Bone marrow (Experimental): core decompression plus autologous concentrated bone marrow
  Interventions: Procedure: core decompression with autologous bone marrow implantation

INTERVENTIONS:
Procedure: core decompression with autologous bone marrow implantation — core biopsy with injection of 40 ml concentrated autologous bone marrow.
  Arms: Bone marrow
Procedure: core decompression of the femoral head — core biopsy with injection of 40 ml saline solution in place of bone marrow.
  Arms: Control

SUMMARY:
In stage 3 Osteonecrosis (ON) of the femoral head, a beneficial effect of bone marrow grafting was reported with a reduction of the functional evolution and the necessity of a total prosthesis placement in a non-controlled retrospective trial. Based on this experience, the investigators would like to start a randomized controlled double blind study on the effect of autologous implantation of autologous bone marrow cells into the necrotic lesion of stage 3 ON of the femoral head.

ELIGIBILITY:
Inclusion Criteria:

1. patients who have a non traumatic ON of the femoral head
2. Stage 3 ON (subchondral fracture).
3. Age > 18 years
4. Be able and willing to participate in the study

Exclusion Criteria:

1. evidence of malignant disorder in the past five years
2. Patient unable to undergo a MRI.
3. Patient who is positive for an HIV, hepatitis B or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
reduction of total prosthesis | 24, 60 months
  Need to undergo a surgical treatment total prosthesis

SECONDARY OUTCOMES:
Pain reduction | 24, 60 months
  Visual analogue scale
functional status | 24, 60 months
  Lequesne and WOMAC scores

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liège, Liège, Liège, Belgium

REFERENCES:
- [Derived] Hauzeur JP, De Maertelaer V, Baudoux E, Malaise M, Beguin Y, Gangji V. Inefficacy of autologous bone marrow concentrate in stage three osteonecrosis: a randomized controlled double-blind trial. Int Orthop. 2018 Jul;42(7):1429-1435. doi: 10.1007/s00264-017-3650-8. Epub 2017 Oct 7. PMID 28988340